CLINICAL TRIAL: NCT05244564
Title: Computer Monitor Versus Augmented Reality: Expanding 3MDR Therapy for PTSD
Brief Title: Computer Monitor vs Augmented Reality 3MDR for PTSD PTSD: A Randomized Controlled Trial
Acronym: CARE4PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Military Traumatic Brain Injury Initiative, USUHS (Unknown); Center for Rehabilitation Sciences Research, USUHS (Unknown)
Responsible Party: Principal Investigator, Michael Roy, Professor of Medicine, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USUHS.2021-076
Record Dates: First submitted 2021-08-11; First posted 2022-02-17 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: All receive the 3MDR intervention, but are randomized to delivery via AR HMD vs via curved high definition gaming computer monitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3MDR delivered via Augmented Reality Head Mounted Display (Experimental): All participants will complete 10-14 treatment sessions (three preparatory sessions, 6 to 10 3MDR therapy sessions, and one concluding session), led by a therapist who has completed training and/or is experienced in the conduct of this form of therapy.
  Interventions: Other: Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR)
- 3MDR delivered via 34-inch curved screen high definition gaming computer monitor (Active Comparator): All participants will complete 10-14 treatment sessions (three preparatory sessions, 6 to 10 3MDR therapy sessions, and one concluding session), led by a therapist who has completed training and/or is experienced in the conduct of this form of therapy.
  Interventions: Other: Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR)

INTERVENTIONS:
Other: Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR) — "Walk and talk" therapy, walking on a treadmill while talking with a therapist about self-chosen pictures representative of one's trauma; 3MDR also includes some features of virtual reality exposure therapy (VRET) and Eye Movement Desensitization and Reprocessing (EMDR) therapy.

SUMMARY:
This is a prospective randomized controlled trial comparing two ways of delivering Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR) therapy for posttraumatic stress disorder (PTSD). The study seeks 60 volunteers who have PTSD and are eligible for care in the Department of Defense healthcare system. There will be 10-14 therapy sessions that are 60-90 minutes long, about once a week, and symptoms will be assessed before and after the therapy as well as 3 and 6 months after completing therapy. 3MDR asks you to choose pictures and music that are integrated into a virtual reality environment. You will be walking on a treadmill throughout each therapy session, while the therapist stands next to the treadmill and asks you questions about the pictures you chose.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) frequently occurs after combat and other life-threatening or traumatic events. Currently available treatments for PTSD often have a brief, limited effect, or are not well-tolerated. Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR) is a new and unique treatment for PTSD that has been commonly referred to as "walk and talk" therapy, because you walk on a treadmill as you work through your symptoms with a therapist. 3MDR also combines some features of virtual reality exposure therapy (VRET) and Eye Movement Desensitization and Reprocessing (EMDR), and has usually been conducted in the Computer Assisted Rehabilitation Environment (CAREN), a sophisticated virtual reality "cave". Previous clinical studies by us and others across several nations have proven the effectiveness of the 3MDR approach in treating symptoms of PTSD. However, the CAREN is large, expensive (~$1 million), and only available in a few places around the world. To try to make 3MDR available to more people, this study will compare how much PTSD symptoms change with 3MDR delivered via two different mechanisms: 1) walking on a regular treadmill while wearing goggles (known as augmented reality head-mounted display, or AR HMD, specifically the Microsoft Hololens2) that allow you to see the treadmill and things around you in the real world, while also seeing pictures in a virtual world, with 2) walking on the same treadmill, with presentation of pictures on a 34-inch curved high definition gaming computer monitor positioned at eye level directly in front of the treadmill. There will be a total of 60 participants in the study, all at Uniformed Services University. After completing the informed consent process, all participants will be evaluated to confirm that they meet criteria for PTSD. There will be two introductory sessions where you meet the therapist you will be working with, and they will help you choose music and pictures that will be used in your later sessions. These introductory sessions can be done in person or virtually. In the third session you will try walking on the treadmill with a sample picture, via either the AR HMD or the computer monitor, depending on which approach you are randomized to receive-you have an equal chance of either. Starting with the 4th session, you will be talking through the pictures you have chosen, with your therapist. You will spend about 10 minutes on each picture, and do 5 or 6 pictures each session, and will do this through session 9. After that, you will complete a brief questionnaire about your symptoms. If you still have significant symptoms, you will do another 2 sessions of talking through your pictures, then do another questionnaire, and again will do two more sessions if you still have symptoms. There is then one final wrap-up session, which can be done either in person or virtually, to discuss how you did with the therapy, and whether you might need any more therapy to help you if you have any symptoms left to address. Depending on how quickly your symptoms improve, you may do a total of 10, 12 or 14 therapy sessions in this study. After you have finished the therapy sessions, you will again be assessed to see how much your symptoms have improved, and you will do this again 3 and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Service member, veteran, retiree, or DEERS-eligible dependent, male or female, at least 18 years or older
* Diagnosis of PTSD, as confirmed by the CAPS-5
* Able to ambulate with contact guard assistance or less, and walk unassisted on a treadmill, at a normal pace, for up to 90 minutes continuously

Exclusion Criteria:

* History of epilepsy or a seizure disorder, other than febrile seizures that occurred during childhood and have not recurred since
* History of a psychotic disorder, bipolar disorder, or active suicidal or homicidal ideation
* Use of benzodiazepines on a regular basis within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD scale for DSM5 (CAPS-5) | 3 months
  The primary outcome measure will be the Clinician Administered PTSD scale for DSM5 (CAPS-5), the gold standard measure for PTSD diagnosis, to assess PTSD symptom severity.
PTSD Checklist for DSM5 (PCL5) | 3 months
  The PTSD Checklist for DSM5 (PCL5), a well-validated 20-item self-report measure of PTSD symptom severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire Depression module (PHQ-9) | 3 months
  The Patient Health Questionnaire Depression module (PHQ-9) is a well-validated instrument for assessing depression symptom severity.
Insomnia Severity Index (ISI) | 3 months
  The Insomnia Severity Index (ISI) is a validated method with which to evaluate insomnia and sleep difficulties.
Neurobehavioral Symptom Inventory (NSI) | 3 months
  The Neurobehavioral Symptom Inventory (NSI) is a validated instrument for assessing postconcussive symptom severity.
Brief Resilience Scale (BRS) | 3 months
  The Brief Resilience Scale (BRS) is a validated instrument used to assess resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roy, MD, MPH, Principal Investigator — Unformed Services University
Locations (1):
- Uniformed Services University, Bethesda, Maryland, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT05244564/ICF_000.pdf